CLINICAL TRIAL: NCT02090660
Title: Feasibility of a Novel Minimally Invasive Technique for Localization of Pulmonary Nodules Using the Spy Thoracoscope System
Brief Title: Technique for Localization of Pulmonary Nodules Using Spy Thoracoscope System
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University Health Network, Toronto (Other)
Collaborators: Novadaq Technologies ULC, now a part of Stryker (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 12-5454
Record Dates: First submitted 2014-03-10; First posted 2014-03-18 (Estimated); Last update posted 2018-02-26 (Actual); Status verified 2018-02

CONDITIONS: Lung Cancer
MeSH Terms: conditions — Lung Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- VATS wedge lung resection (Experimental)
  Interventions: Other: ICG Localization with Spy thoracoscope localization

INTERVENTIONS:
Other: ICG Localization with Spy thoracoscope localization

SUMMARY:
This study will determine the feasibility of the novel Indocyanine Green (ICG) fluorescence localization technique with a Laser fluorescence thoracoscope system.

The primary objective of this study is to prove the validity and safety of our novel fluorescent localization method with utilized ICG and novel near infra-red fluorescence videoscope system.

ELIGIBILITY:
Inclusion Criteria:

* Any patient scheduled for a VATS wedge lung resection using CT guided micro-coil lung implantation for the localization of the lung lesion.

Exclusion Criteria:

* Any patients with an allergy to iodine, shellfish, or cough mixture, betadine or other iodine contrast agents.
* Pregnant or potentially pregnant women.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2014-04; Primary Completion 2016-02 (Actual)

PRIMARY OUTCOMES:
Compare incidence of Adverse Events (AE) occurrence due to ICG injection with micro-coil placement versus overall AE occurrence for micro-coil placement alone. | Within 4 hours of ICG injection

CONTACTS AND LOCATIONS:
Overall Officials: Kazuhiro Yasufuku, MD, Principal Investigator — University Health Network, Toronto
Locations (1):
- University Health Network: Toronto General Hospital, Toronto, Ontario, Canada